CLINICAL TRIAL: NCT06309394
Title: An Open-Label Study Assessing the Mass Balance, Pharmacokinetics, and Metabolite Profiles of a Single Oral Dose of [14C]INCB099280 in Healthy Male Participants
Brief Title: A Study Assessing the Mass Balance, Pharmacokinetics, and Metabolite Profiles of a Single Oral Dose of [14C]INCB099280 in Healthy Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: INCB99280-102
Record Dates: First submitted 2024-02-23; First posted 2024-03-13 (Actual); Results first posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-08

CONDITIONS: Healthy Participants
Keywords: INCB099280

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- INCB099280 (Experimental): Participants will be administered INCB099280 tablet orally, followed approximately 10 minutes later by an oral dose solution of radiolabeled INCB099280.
  Interventions: Drug: INCB099280

INTERVENTIONS:
Drug: INCB099280 — INCB099280 will be administered orally, followed approximately 10 minutes later by an oral dose solution of radiolabeled INCB099280.

SUMMARY:
This study is being conducted to assess the Mass Balance, Pharmacokinetics, and Metabolite Profiles of a Single Oral Dose of [14C]INCB099280 in Healthy Male Participants.

ELIGIBILITY:
Inclusion Criteria:

* Ability to comprehend and willingness to sign a written ICF for the study.
* Healthy males, as determined by the investigator based upon physical examinations, ECGs, vital signs, and safety laboratory assessments, aged 35 to 55 years, inclusive, at the time of signing the ICF.
* Body mass index between 18.0 and 32.0 kg/m2, inclusive, at the time of screening.
* No clinically significant findings in screening evaluations (eg, clinical, laboratory, vital signs, and ECG) at screening and Day -1.
* Ability to swallow and retain oral medication.

Exclusion Criteria:

* History of clinically significant respiratory, renal, gastrointestinal, endocrine, hematopoietic, psychiatric, and/or neurological disease as judged by the investigator.
* History of cardiovascular, cerebrovascular, peripheral vascular, or thrombotic disease or uncontrolled hypertension (systolic blood pressure > 140 mm Hg or diastolic blood pressure > 90 mmHg at screening, confirmed by repeat testing).
* Presence of a malabsorption syndrome (eg, Crohn's disease or chronic pancreatitis) that could possibly affect drug absorption.
* Current or recent (within 6 months before screening), clinically significant, gastrointestinal disease or surgery (including cholecystectomy, excluding appendectomy) that could affect the absorption of study drug.
* Any major surgery within 6 months of screening.
* Donation of blood to a blood bank or in a clinical study (except a screening visit) within 3 months before screening (within 2 weeks for plasma donation).
* Positive test for HBV, HCV, or HIV at screening. Participants whose HBV results are compatible with prior immunization or immunity due to infection may be included at the discretion of the investigator.
* Regular alcohol consumption > 21 units per week (1 unit = 8 oz of beer or a 25-mL shot of a 40% spirit; 1.5 to 2 units = a 125-mL glass of wine, depending on type).
* Positive breath test for alcohol or positive urine screen for drugs of abuse (confirmed by repeat) at screening or admission (Day -1).
* Treatment with another investigational medication within 90 days or 5 half-lives (whichever is longer) before Day 1 or current enrollment in another investigational drug study.
* Participation in any clinical study involving a 14C-radiolabeled investigational product within 12 months prior to admission (Day -1).
* Radiation exposure, including that from the present study, excluding background radiation but including diagnostic x-rays and other medical exposures, exceeding 5 mSv in the last 12 months or 10 mSv in the last 5 years. No occupationally exposed worker, as defined in the Ionising Radiation Regulations 2017, shall participate in the study.
* History of tobacco- or nicotine-containing product use within 1 month before screening. Consumption of tobacco- or nicotine-containing products 72 hours before admission (Day -1) until CRU discharge is not permitted. Breath test for carbon monoxide > 10 ppm (confirmed by repeat) at screening or admission (Day -1).
* Use of prescription drugs within 14 days before Day 1 or nonprescription medications/products (including vitamins, minerals, and phytotherapeutic, herbal, or plant-derived preparations) within 7 days before Day 1 until CRU discharge. However, paracetamol up to 4000 mg Q24H and ibuprofen up to 600 mg Q24H are permitted.

Other protocol-defined Inclusion/Exclusion Criteria may apply.

Ages: 35 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Incyte Medical, Study Director — Incyte Corporation
Locations (1):
- Quotient Sciences Ltd, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- INCB099280 400 mg + [14C]INCB099280 78.3 μCi: Participants received a single dose of INCB099280 400 milligrams (mg) administered in tablet form (4 × 100-mg tablets) followed approximately 10 minutes later by an oral dose solution containing 78.3 microcuries (μCi) (2.9 megabecquerel [MBq]) of [14C]INCB099280 (not more than 97.2 μCi [3.6 MBq]).
Period: Overall Study
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (5.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Total Recovery (Urine + Feces) of the Administered Radioactivity
Description: Radioactivity in urine and feces was reported as the percentage of the administered radioactivity excreted.
Time Frame: 264 hours in urine; 408 hours in feces
Population: Pharmacokinetic (PK)-Evaluable Population: all participants who received the study treatment and provided at least 1 postdose PK sample.
Measure: Median (Full Range); unit: percentage of radioactivity
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
percentage of radioactivity | 83.2 [78.3 to 89.5]

2. Secondary Outcome: Abundance of INCB099280 Detected in Plasma
Description: Plasma samples for metabolism investigations were obtained at 0, 1, 2, 4, 8, 12, 16, and 24 hours post-dose and were pooled across participants at each timepoint. TRPA=total radioactive peak area. The reported values are single measurements of pooled plasma or fecal samples; therefore, no statistical analysis is possible, and data have been reported with a measure type of "number."
Time Frame: 0 hours (predose) and up to 24 hours post-dose
Population: PK-Evaluable Population
Measure: Number; unit: percentage of TRPA
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
percentage of TRPA
  1 hour post-dose | 33.4
  2 hours post-dose | 70.3
  4 hours post-dose | 57.2
  8 hours post-dose | 35.3
  12 hours post-dose | 38.3
  16 hours post-dose | 44.9
  24 hours post-dose | 23.2

3. Secondary Outcome: Abundance of INCB099280 Metabolites Detected in Feces
Description: Homogenized fecal samples from individual participants were pooled for each collection interval by taking a fixed percentage of the total amount excreted from each collection interval/participant. The reported values are single measurements of pooled plasma or fecal samples; therefore, no statistical analysis is possible, and data have been reported with a measure type of "number."
Time Frame: 0 hours (predose) and up to 96 hours post-dose
Population: PK-Evaluable Population
Measure: Number; unit: percentage of total dosed radioactivity
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
percentage of total dosed radioactivity
  INCB099280, 0 to 24 hours post-dose | 1.98
  INCB099280, 24 to 48 hours post-dose | 13.3
  INCB099280, 48 to 72 hours post-dose | 36.6
  INCB099280, 72 to 96 hours post-dose | 5.37
  M12, 0 to 24 hours post-dose | 0
  M12, 24 to 48 hours post-dose | 2.30
  M12, 48 to 72 hours post-dose | 4.06
  M12, 72 to 96 hours post-dose | 1.63

4. Secondary Outcome: Cmax of INCB099280
Description: Cmax was defined as the maximum observed plasma or serum concentration of INCB099280.
Time Frame: 0 hours (predose) and 0.5, 1, 2, 4, 6, 8, 12, and 16 hours post-dose (Day 1); 24 and 36 hours post-dose (Day 2); 48 hours post-dose (Day 3), 72 hours post-dose (Day 4), 96 hours post-dose (Day 5), 120 hours post-dose (Day 6)
Population: PK-Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomolar
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
nanomolar | 994 (90.8)

5. Secondary Outcome: Tmax of INCB099280
Description: tmax was defined as the time to the maximum concentration of INCB099280.
Time Frame: as for outcome 4
Population: PK-Evaluable Population
Measure: Median (Full Range); unit: hours
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
hours | 4.0 [2.0 to 4.2]

6. Secondary Outcome: AUC0-t of INCB099280
Description: AUC0-t was defined as the area under the steady-state plasma or serum concentration-time curve up to the last measurable concentration of INCB099280.
Time Frame: as for outcome 4
Population: PK-Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours * nanomolar
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
hours * nanomolar | 11100 (118)

7. Secondary Outcome: AUC0-∞ of INCB099280
Description: AUC0-∞ was defined as the area under the single-dose plasma or serum concentration-time curve extrapolated to time of infinity.
Time Frame: as for outcome 4
Population: PK-Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours * nanomolar
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
hours * nanomolar | 11200 (117)

8. Secondary Outcome: t½ of INCB099280
Description: t½ was defined as the apparent terminal-phase disposition half-life of INCB099280.
Time Frame: as for outcome 4
Population: PK-Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
hours | 14.8 (17.9)

9. Secondary Outcome: CL/F of INCB099280
Description: CL/F was defined as the apparent oral dose clearance of INCB099280.
Time Frame: as for outcome 4
Population: PK-Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
liters per hour | 46.9 (117)

10. Secondary Outcome: Vz/F of INCB099280
Description: Vz/F was defined as the maximum observed plasma or serum concentration of INCB099280.
Time Frame: as for outcome 4
Population: PK-Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
liters | 1000 (91.3)

11. Secondary Outcome: Cmax of Total Radioactivity in Blood
Description: Cmax was defined as the maximum observed concentration of total radioactivity in blood. Additional samples were collected every 24 hours until discharge (up to 264 hours).
Time Frame: as for outcome 4
Population: PK-Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomolar
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
nanomolar | 1010 (61.1)

12. Secondary Outcome: Tmax of Total Radioactivity in Blood
Description: tmax was defined as the time to the maximum concentration of total radioactivity in blood. Additional samples were collected every 24 hours until discharge (up to 264 hours).
Time Frame: as for outcome 4
Population: PK-Evaluable Population
Measure: Median (Full Range); unit: hours
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
hours | 4.0 [2.0 to 4.2]

13. Secondary Outcome: AUC0-t of Total Radioactivity in Blood
Description: AUC0-t was defined as the area under the steady-state plasma or serum concentration-time curve up to the last measurable concentration of total radioactivity in blood. Additional samples were collected every 24 hours until discharge (up to 264 hours).
Time Frame: as for outcome 4
Population: PK-Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours * nanomolar
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
hours * nanomolar | 14100 (79.5)

14. Secondary Outcome: AUC0-∞ of Total Radioactivity in Blood
Description: AUC0-∞ was defined as the area under the single-dose plasma or serum concentration-time curve extrapolated to time of infinity. Additional samples were collected every 24 hours until discharge (up to 264 hours).
Time Frame: as for outcome 4
Population: PK-Evaluable Population. Analysis was not conducted as %AUCextrapolation ≥ 20%.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours * nanomolar
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
hours * nanomolar | 37200 (151)

15. Secondary Outcome: t½ of Total Radioactivity in Blood
Description: t½ was defined as the apparent terminal-phase disposition half-life of total radioactivity in blood. Additional samples were collected every 24 hours until discharge (up to 264 hours).
Time Frame: as for outcome 4
Population: PK-Evaluable Population. Analysis was not conducted as Rsq_adjusted ≤ 0.7 and/or %AUCextrapolation ≥ 20%.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
hours | 36.1 (321)

16. Secondary Outcome: CL/F of Total Radioactivity in Blood
Description: CL/F was defined as the apparent oral dose clearance of total radioactivity in blood. Additional samples were collected every 24 hours until discharge (up to 264 hours).
Time Frame: as for outcome 4
Population: PK-Evaluable Population. Analysis was not conducted as %AUCextrapolation ≥ 20%.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
liters per hour | 14.2 (151)

17. Secondary Outcome: Vz/F of Total Radioactivity in Blood
Description: Vz/F was defined as the maximum observed plasma or serum concentration of total radioactivity in blood. Additional samples were collected every 24 hours until discharge (up to 264 hours).
Time Frame: as for outcome 4
Population: PK-Evaluable Population. Analysis was not conducted as %AUCextrapolation ≥ 20%.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
liters | 738 (69.7)

18. Secondary Outcome: Cmax of Total Radioactivity in Plasma
Description: Cmax was defined as the maximum observed concentration of total radioactivity in plasma. Additional samples were collected every 24 hours until discharge (up to 264 hours).
Time Frame: as for outcome 4
Population: PK-Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomolar
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
nanomolar | 1450 (69.3)

19. Secondary Outcome: Tmax of Total Radioactivity in Plasma
Description: tmax was defined as the time to the maximum concentration of total radioactivity in plasma. Additional samples were collected every 24 hours until discharge (up to 264 hours).
Time Frame: as for outcome 4
Population: PK-Evaluable Population
Measure: Median (Full Range); unit: hours
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
hours | 4.0 [2.0 to 4.2]

20. Secondary Outcome: AUC0-t of Total Radioactivity in Plasma
Description: AUC0-t was defined as the area under the steady-state plasma or serum concentration-time curve up to the last measurable concentration of total radioactivity in plasma. Additional samples were collected every 24 hours until discharge (up to 264 hours).
Time Frame: as for outcome 4
Population: PK-Evaluable Population
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours * nanomolar
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
hours * nanomolar | 14100 (126)

21. Secondary Outcome: AUC0-∞ of Total Radioactivity in Plasma
Description: as for outcome 14
Time Frame: as for outcome 4
Population: PK-Evaluable Population. Only participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours * nanomolar
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
hours * nanomolar | 18500 (105)

22. Secondary Outcome: t½ of Total Radioactivity in Plasma
Description: t½ was defined as the apparent terminal-phase disposition half-life of total radioactivity in plasma. Additional samples were collected every 24 hours until discharge (up to 264 hours).
Time Frame: as for outcome 4
Population: PK-Evaluable Population. Only participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
hours | 8.88 (57.6)

23. Secondary Outcome: CL/F of Total Radioactivity in Plasma
Description: CL/F was defined as the apparent oral dose clearance of total radioactivity in plasma. Additional samples were collected every 24 hours until discharge (up to 264 hours).
Time Frame: as for outcome 4
Population: PK-Evaluable Population. Only participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters per hour
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
liters per hour | 28.5 (105)

24. Secondary Outcome: Vz/F of Total Radioactivity in Plasma
Description: Vz/F was defined as the maximum observed plasma or serum concentration of total radioactivity in plasma. Additional samples were collected every 24 hours until discharge (up to 264 hours).
Time Frame: as for outcome 4
Population: PK-Evaluable Population. Only participants with available data were analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
liters | 365 (40.4)

25. Secondary Outcome: Number of Participants With Any Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not it was considered drug-related. An AE could be any unfavorable or unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of study treatment. A TEAE was defined as any AE either reported for the first time or the worsening of a pre-existing event after the first dose of study drug.
Time Frame: up to Day 22
Population: Safety Population: all participants who received the study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
Number analyzed (Participants) | 5
Participants | 1

ADVERSE EVENTS:
Time Frame: from signing of the Informed Consent Form until up to Day 22
Description: Adverse events were analyzed in the Safety Population, comprised of all participants who received the study treatment.
Arm/Group | INCB099280 400 mg + [14C]INCB099280 78.3 μCi
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | INCB099280 400 mg + [14C]INCB099280 78.3 μCi (N=5)
Diarrhoea (Gastrointestinal disorders) | 1
Anxiety (Psychiatric disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Following the first publication, the Institution and/or Principal Investigator may publish data or results from the Study, provided, however, that the Institution and/or Principal Investigator submits the proposed publication to the Sponsor for review at least sixty (60) days prior to the date of the proposed publication. Sponsor may remove from the proposed publication any information that is considered confidential and/or proprietary other than Study data and results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-25): https://cdn.clinicaltrials.gov/large-docs/94/NCT06309394/Prot_SAP_000.pdf